CLINICAL TRIAL: NCT01044732
Title: Third Eye Retroscope Randomized Clinical Evaluation (The "TERRACE" Study)
Brief Title: Third Eye Retroscope Randomized Clinical Evaluation
Acronym: TERRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avantis Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Avantis TER-08-06
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Results first posted 2015-10-01 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal; Neoplasms; Adenomas; Polyps; Miss rates; Detection rates; Colonoscope; Third Eye Retroscope
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Adenoma; Polyps

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - COLO, then TER (Experimental): Complete examination with standard colonoscope ("COLO") followed by complete examination with Third Eye Retroscope ("TER") used in conjunction with standard colonoscope
  Interventions: Device: Third Eye Retroscope
- Group B - TER, then COLO (Active Comparator): Complete examination with Third Eye Retroscope ("TER") used in conjunction with standard colonoscope, followed by complete examination with standard colonoscope ("COLO") alone
  Interventions: Device: Third Eye Retroscope

INTERVENTIONS:
Device: Third Eye Retroscope — Device used with colonoscope to provide second, retrograde view of the colon

SUMMARY:
The Third Eye® Retroscope® is a device that can be inserted through the instrument channel of a standard colonoscope to provide an additional, retrograde (or backward) view that reveals areas behind folds and flexures in the colon, and might detect additional polyps that cannot be seen with the colonoscope alone.

Patients who participate as subjects in the study will undergo two complete colonoscopy procedures, a standard colonoscopy and a colonoscopy in which a Third Eye Retroscope is used along with the same colonoscope. Half of the patients will have the standard colonoscopy first followed by the Third Eye colonoscopy, and the other half will have the Third Eye procedure first.

Results from the two groups will be analyzed and compared to determine the effectiveness of the Third Eye Retroscope for detecting additional adenomas and other polyps compared with the standard colonoscope alone.

DETAILED DESCRIPTION:
Colonoscopy is generally agreed to be the best method for detecting and removing pre-cancerous polyps, but some lesions can be missed, especially if they are located behind folds in the lining of the colon or behind flexures (sharp bends) in the colon.

The Third Eye® Retroscope® is a device that can be inserted through the instrument channel of a standard colonoscope to provide an additional, retrograde (or backward) view that reveals areas behind folds and flexures in the colon. Previous studies have shown the device to be effective for detecting additional polyps that could not have been seen with the colonoscope alone.

The purpose of this research is to compare the additional diagnostic yield obtained by using the Third Eye® Retroscope® vs. the diagnostic yield for the standard colonoscope alone in the context of a randomized, controlled study design.

Patients who are scheduled for colonoscopy will be recruited to the study and randomized to one of two groups. Each patient will undergo two "back-to-back" procedures.

Patients in Group A (study group) will undergo a standard colonoscopy followed immediately by a Third Eye colonoscopy.

Patients in Group B (control group) will undergo a Third Eye colonoscopy followed immediately by a standard colonoscopy.

Results from the two groups will be analyzed and compared to determine the effectiveness of the Third Eye Retroscope for detecting additional adenomas and other polyps compared with the standard colonoscope alone.

ELIGIBILITY:
Inclusion Criteria:

* The patient is undergoing colonoscopy for screening, for surveillance in follow-up of previous polypectomy or for diagnostic workup;
* The patient must understand and provide written consent for the procedure.

Exclusion Criteria:

* Patients with a history of colonic resection;
* Patients with inflammatory bowel disease;
* Patients with a personal history of polyposis syndrome;
* Patients with suspected chronic stricture potentially precluding complete colonoscopy;
* Patients with diverticulitis or toxic megacolon;
* Patients with a history of radiation therapy to abdomen or pelvis;
* Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter D. Siersema, MD, PhD, Principal Investigator — UMC Utrecht
Locations (9):
- United States (5):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Kansas City Veterans Administration Medical Center, Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Bayside Endoscopy Center, Providence, Rhode Island
  - Baylor University Medical Center, Dallas, Texas
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Istituto Clinico Humanitas, Milan, Italy
- University Medical Center Utrecht, Utrecht, Netherlands
- St. Mark's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Aggregated, de-identified data to be published in peer-reviewed medical journal

REFERENCES:
- [Result] Leufkens AM, DeMarco DC, Rastogi A, Akerman PA, Azzouzi K, Rothstein RI, Vleggaar FP, Repici A, Rando G, Okolo PI, Dewit O, Ignjatovic A, Odstrcil E, East J, Deprez PH, Saunders BP, Kalloo AN, Creel B, Singh V, Lennon AM, Siersema PD; Third Eye Retroscope Randomized Clinical Evaluation [TERRACE] Study Group. Effect of a retrograde-viewing device on adenoma detection rate during colonoscopy: the TERRACE study. Gastrointest Endosc. 2011 Mar;73(3):480-9. doi: 10.1016/j.gie.2010.09.004. Epub 2010 Nov 10. PMID 21067735
- [Result] Siersema PD, Rastogi A, Leufkens AM, Akerman PA, Azzouzi K, Rothstein RI, Vleggaar FP, Repici A, Rando G, Okolo PI, Dewit O, Ignjatovic A, Odstrcil E, East J, Deprez PH, Saunders BP, Kalloo AN, Creel B, Singh V, Lennon AM, DeMarco DC. Retrograde-viewing device improves adenoma detection rate in colonoscopies for surveillance and diagnostic workup. World J Gastroenterol. 2012 Jul 14;18(26):3400-8. doi: 10.3748/wjg.v18.i26.3400. PMID 22807609

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A - SC Followed by TEC: Standard colonoscopy (SC) followed by Third Eye colonoscopy (TEC)
  Third Eye colonoscopy: Examination of the colon with a Third Eye Retroscope used in combination with a colonoscope to provide second, retrograde view of the colon
- Group B - TEC Followed by SC: Third Eye colonoscopy (TEC) followed by standard colonoscopy (SC)
  Third Eye colonoscopy: Examination of the colon with a Third Eye Retroscope used in combination with a colonoscope to provide second, retrograde view of the colon
Period: Overall Study
Arm/Group | Group A - SC Followed by TEC | Group B - TEC Followed by SC
Started | 222 | 226
Completed | 173 | 176
Not Completed | 49 | 50
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 5 | 3
Not completed — Protocol Violation | 11 | 12
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Inadequate bowel preparation | 11 | 17
Not completed — Inability to reach cecum | 5 | 2
Not completed — Technical error or malfunction | 15 | 14

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population, i.e., those who were actually examined during the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - SC Followed by TEC | Group B - TEC Followed by SC | Total
Number analyzed (Participants) | 184 | 188 | 372
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (9.8) | 58.0 (9.7) | 57.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 59 | 128
  Male | 115 | 129 | 244
Region of Enrollment [Number; unit: participants in ITT population]
  Netherlands | 19 | 22 | 41
  Belgium | 24 | 26 | 50
  United States | 114 | 111 | 225
  Italy | 25 | 28 | 53
  United Kingdom | 2 | 1 | 3
Indication for colonoscopy procedure [Number; unit: participants in ITT population]
  Screening | 97 | 92 | 189
  Surveillance | 41 | 55 | 96
  Diagnostic | 46 | 41 | 87

OUTCOME MEASURES:

1. Primary Outcome: Detection Rates for Adenomas and for Total Polyps
Description: Numbers of polyps and adenomas detected in first and second procedures for each group
Time Frame: Acute - subjects were followed for the duration of the procedures, an average of 40 minutes.
Population: Per-protocol population
Measure: Number; unit: Polyps or adenomas detected
Arm/Group | Group A - SC Followed by TEC | Group B - TEC Followed by SC
Number analyzed (Participants) | 173 | 176
Polyps or adenomas detected
  Polyps detected in first procedure | 160 | 163
  Polyps detected in second procedure | 78 | 31
  Adenomas detected in first procedure | 107 | 115
  Adenomas detected in second procedure | 49 | 26

2. Secondary Outcome: Times for Withdrawal Phase and for Complete Procedure
Description: For all examinations with each method (SC or TEC), mean time for withdrawal phase and mean time for total procedure
Time Frame: Acute - subjects were followed for the duration of the procedures, an average of 40 minutes.
Population: All subjects in study (i.e., Group A and Group B combined)
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- All SC Procedures: For all subjects in study (i.e., Group A and Group B combined), mean times for withdrawal phase and for total procedure during standard colonoscopies (SC)
- All TEC Procedures: For all subjects in study (i.e., Group A and Group B combined), mean times for withdrawal phase and for total procedure during Third Eye colonoscopies (TEC)
Arm/Group | All SC Procedures | All TEC Procedures
Number analyzed (Participants) | 349 | 349
Minutes
  Mean withdrawal time | 7.58 (2.79) | 9.52 (6.15)
  Mean total procedure time | 16.97 (9.90) | 20.87 (10.06)

ADVERSE EVENTS:
Time Frame: 24-72 hours post-procedure
Description: Assessed through follow-up telephone interview
Arm/Group | Group A - SC Followed by TEC | Group B - TEC Followed by SC
Serious Adverse Events (participants affected / at risk) | 0/184 | 0/188
Other Adverse Events (participants affected / at risk) | 0/184 | 0/188

LIMITATIONS AND CAVEATS:
With mean subject age of 57.8 years, population was younger than in some studies, so polyp prevalence might be below average.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No